CLINICAL TRIAL: NCT01869179
Title: Community Choirs To Promote Healthy Aging And Independence Of Older Adults
Brief Title: Community Choirs To Promote Healthy Aging; Community of Voices Chorus
Acronym: COV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco Community Music Center (Unknown); Department of Aging and Adults Services San Francisco (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R01AG042526 (NIH)
Record Dates: First submitted 2013-01-09; First posted 2013-06-05 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Well Being
Keywords: Well being; Low income; Choir singing; Spanish speaking; Community based; Seniors; 60+ aged adults; health disparities

STUDY DESIGN:
Intervention Model Description: Cluster-randomized controlled design
Masking Description: Randomization assignment was not revealed to study personnel or study participants until after baseline assessments were completed for each pair of centers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community of Voices choir program (Experimental): Participants will receive the 12 month choir program as soon as possible after study enrollment.
  Interventions: Behavioral: Community of Voices choir program
- Wait-list control group (Experimental): Waits six months, and at the end of the six months is offered the option of participating in the 12 month choir program.
  Interventions: Behavioral: Community of Voices choir program; Behavioral: Wait-list control group

INTERVENTIONS:
Behavioral: Community of Voices choir program — Attend weekly choir sessions for 12 months at the Senior Center. All choir sessions will include activities that focus on cognitive, psychosocial, and physical engagement components Choir sessions will last 90 minutes each with a 10 minute break. Take part in 3-4 informal choir concerts.
Behavioral: Wait-list control group
  Arms: Wait-list control group

SUMMARY:
The investigators will recruit 450 older adults and will utilize 12 Administration on Aging (AoA)-supported senior centers to implement a multisite, cluster randomized (by center), wait-list clinical trial. Centers will be randomized to receive the choir program immediately (intervention group) or after a 6-month delayed intervention phase (control group). The community choirs will be led by professional music directors. The investigators will assess both primary and secondary outcomes at baseline, 6 and 12 months, with the main intervention group comparison being at 6 months. The investigators will also evaluate the start-up and ongoing program costs for senior centers, including cost/person served and determine quality adjusted life years.

The hypotheses are:

1. Compared to delayed intervention controls, participation in a community choir program will be associated with improvements/maintenance on the primary outcomes of physical function (balance, walking speed, strength), depressive symptoms, and cognition (executive function and memory) at 6 months. The investigators also predict within-group improvements on these primary outcomes at 12 months.
2. Compared to delayed intervention controls, participation in a community choir program will be associated with improvements in the secondary outcomes of well-being (depressive symptoms, loneliness, resilience, social participation, health-related quality of life, shortness of breath, functional status, falls, and health services use) at 6 months. The investigators also predict within-group improvements on these secondary outcomes at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 and older
* Living independently
* Have adequate visual and auditory acuity (with correction) to complete testing
* Speak English or Spanish (including both bilingual and monolingual Spanish speakers)

Exclusion Criteria:

* A baseline diagnosis of dementia, determined by the screening tool or self-report of diagnosis
* Have an unstable or serious medical condition that would limit participation in the weekly choir sessions or assessments, including current (but not prior) severe psychiatric disorder
* Currently singing in a choir, within the last 6 months
* Plans to move out of the area within 12 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Physical function | up to 12 months
  We will measure several physical function outcomes. The Short Physical Performance Battery (SPPB) chair stands will be the primary outcome measure. Baseline, 6 months, 12 months. Additional motor function outcomes using the NIH Toolbox are listed below.
Cognitive Function | up to 12 months
  We will use the Trailmaking Test as a primary outcome of executive function. Baseline, 6 months, 12 months. Additional tests of executive function and memory are listed as secondary outcomes.
Depressive Symptoms | up to 12 months
  We will use the Patient Health Questionnaire (PHQ-8) as a primary measure of depressive symptoms. Baseline, 6 months, 12 months. Additional NIH Toolbox Emotion measures are listed as secondary outcomes.

SECONDARY OUTCOMES:
Health-Related Quality of Life | up to 12 months
  We will use the brief, self-report European Quality of Life (EQ-5D) to measure health-related quality of life. It has versions in both English and Spanish and also alternate and phone versions. It covers five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Baseline, 6 months, 12 months
Health Care Services Utilization | up to 12 months
  We will track utilization of health care services for cost analysis. The list of health care services is modified from the Chronic Disease Self-Management study and includes visits to a doctor, mental health provider (e.g., counselor, psychologist), other health providers (e.g., home health nurse, physical therapist), and emergency room and hospitalizations (and reason for stay). Participants (including those on the wait-list) will be contacted by phone every three months to complete the form about health care services used in the prior three months. Baseline, 6 months, 12 months
Falls | up to 12 months
  We will query frequency of falls using a single question commonly used in several large diverse studies about falls. Falls will also be assessed by phone every three months. Baseline, 6 months, 12 months
Shortness of breath | up to 12 months
  We will ask three questions about shortness of breath based on Blazer and colleagues. Baseline, 6 months, 12 months
Balance and Endurance | up to 12 months
  We will use the NIH Toolbox Motor to assess endurance (4 Meter Walk Gait Speed Test) and balance (Standing Balance Test). Baseline, 6 months, 12 months.
Memory and Executive Function | up to 12 months
  As secondary cognitive outcomes, we will use the NIH Toolbox to assess executive function and attention (NIH Toolbox Flanker Inhibitory Control and Attention Test) and verbal memory (NIH Toolbox Auditory Verbal Learning Test - Rey). Baseline, 6 months, 12 months.
Emotion | up to 12 months
  We will also be using the NIH Toolbox to assess additional aspects of emotion, including psychological well-being (Positive Affect), Self-Efficacy, social relationships (Emotional Support, Friendship, Loneliness), negative affect (Fear-Affect, Sadness), Medical Outcomes Study (MOS) social support, and Apathy. Baseline, 6 months, 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Julene K Johnson, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Institute for Health & Aging, San Francisco, California, United States

REFERENCES:
- [Background] Johnson JK, Napoles AM, Stewart AL, Max WB, Santoyo-Olsson J, Freyre R, Allison TA, Gregorich SE. Study protocol for a cluster randomized trial of the Community of Voices choir intervention to promote the health and well-being of diverse older adults. BMC Public Health. 2015 Oct 13;15:1049. doi: 10.1186/s12889-015-2395-9. PMID 26463176
- [Result] Johnson JK, Gregorich SE, Acree M, Napoles AM, Flatt JD, Pounds D, Pabst A, Stewart AL. Recruitment and baseline characteristics of the Community of Voices choir study to promote the health and well-being of diverse older adults. Contemp Clin Trials Commun. 2017 Dec;8:106-113. doi: 10.1016/j.conctc.2017.09.006. Epub 2017 Sep 17. PMID 29399643
- [Result] Johnson JK, Stewart AL, Acree M, Napoles AM, Flatt JD, Max WB, Gregorich SE. A Community Choir Intervention to Promote Well-Being Among Diverse Older Adults: Results From the Community of Voices Trial. J Gerontol B Psychol Sci Soc Sci. 2020 Feb 14;75(3):549-559. doi: 10.1093/geronb/gby132. PMID 30412233
- [Derived] Allison TA, Napoles AM, Johnson JK, Stewart AL, Rodriguez-Salazar M, Peringer J, Sherman S, Ortez-Alfaro J, Villero O, Portacolone E. Multi-cultural perspectives on group singing among diverse older adults. Geriatr Nurs. 2020 Nov-Dec;41(6):1006-1012. doi: 10.1016/j.gerinurse.2020.07.011. Epub 2020 Aug 8. PMID 32778434
- See also: Community of Voices trial website, including program manual — https://cov.ucsf.edu/